CLINICAL TRIAL: NCT05818241
Title: Study on the Immediate Recovery and Satisfaction After Distal Radius Fracture During the First Three Months- a PROM Based Observational Study With Day-to-day Records
Brief Title: Satisfaction and Recovery After Distal Radius Fracture
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Joakim Stromberg, senior consultant,, Sahlgrenska University Hospital
Other Study IDs: DRFx STAR
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Distal Radius Fracture
Keywords: wrist function; recovery
MeSH Terms: conditions — Wrist Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cast: Patients that are conservatively treated (in a cast, either without or with reduction)
  Interventions: Procedure: Surgical treatment of fracture
- Surgery: Patients that undergo surgical treatment (regardless of method)
  Interventions: Procedure: Treatment of fracture by forearm cast

INTERVENTIONS:
Procedure: Treatment of fracture by forearm cast — Patient that are not surgically treated for DRF
  Other Names: casting, conservative treatment
  Groups: Surgery
Procedure: Surgical treatment of fracture — Patients that are surgically treated for DRF
  Groups: Cast

SUMMARY:
Distal radius fracture is the most common fracture in Sweden, but little is known about the patient's experience of pain and hand function during the first three months after the injury. This observational study will provide detailed information on a daily basis regarding pain, use of analgesic drugs, use of splints and hand function as measured weekly by a condition-specific questionnaire.

DETAILED DESCRIPTION:
Two hundred patients who are treated conservatively in a cast and one hundred patients who have undergone surgery will be asked to complete a questionnaire with the following outcome measures for three months:

1. Pain (day-by-day registration on a Likert scale, range 0-10)
2. Analgesic used (day-by-day registration of specific drug, dose and number)
3. PRWE (Patient Reported Wrist Evaluation form, week-by-week registration)
4. Use of and evaluation of efficacy of prefabricated wrist splints (week-by-week registration)
5. Details of sick leave and return to work at completion of the questionnaire at three months.

The study is entirely PROM-based and the patient will not require any additional appointments.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral distal radius fractures in patients without any other significant injuries regardless of ligament injuries and ulnar fractures.
* Signed written consent

Exclusion Criteria:

* Compound injuries
* Open fractures
* Patients with post traumatic function deficits at any level in the affected arm prior to the distal radius fracture.
* Patients with function deficits in the affected arm due to other medical conditions (e.g. Parkinsons disease, Rheumatoid Arthritis)
* Reduced mental capacity (e.g. dementia, substance abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a distal radius fracture with the inclusion criteria and without the exclusion criteria at the emergency ward are eligible .
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported hand function | Every week for three months
  Patient Rated Wrist Evaluation (PRWE) questionnaire

SECONDARY OUTCOMES:
Day-by-day pain record | Every day for three months
  Patient reported pain as measured on a Likert scale 0-10 (0=no pain, 10= maximum pain)
Analgesics | Every day for three months
  Daily record of use of analgesic drugs
Wrist splint usage | Every week for three months
  Patient reported use of splint and evaluation of its efficacy

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Department of Hand Therapy, Mölndal, Region Västra Götaland
  - Alingsås Lasarett/ District Hospital, Alingsås